CLINICAL TRIAL: NCT06592560
Title: Diagnostic Value of Asprosin As a Biomarker in Breast Cancer
Brief Title: Asprosin in Breast Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Marina Hanna Thabet Ghobrial (Other)
Responsible Party: Sponsor-Investigator, Marina Hanna Thabet Ghobrial, Assistant Lecturer, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Asprosin
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Enzyme-Linked Immunosorbent Assay

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Healthy people
  Interventions: Device: ELISA
- Patients with benign breast lesions
  Interventions: Device: ELISA
- Patients with breast cancer
  Interventions: Device: ELISA

INTERVENTIONS:
Device: ELISA — Specific test: Assay of asprosin marker will be measured by enzyme-linked immunosorbent assay ( ELISA).

SUMMARY:
To evaluate the clinical utility of Asprosin measurement in breast cancer patients in comparison with healthy controls and patients with benign breast lesions.

To compare between Asprosin and the routine markers (CEA, CA15-3) as biomarkers for breast cancer diagnosis

ELIGIBILITY:
Inclusion Criteria:

-

Females aged (40 ± 20 years) who did not receive any chemotherapy or surgical treatment and they will be divided as follow:

Group 1: healthy controls from healthy volunteers. Group 2: patients with benign breast lesions. Group 3: breast cancer patients.

Exclusion Criteria:

* 1- Female patients with any other type of malignant or benign tumors. 2- Past history of chemotherapy or surgical treatment of cancer.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Group 1: healthy controls from healthy volunteers. Group 2: patients with benign breast lesions. Group 3: breast cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Diagnostic value of Asprosin as a biomarker in breast cancer | Baseline
  Evaluation of the clinical utility of measurement of asprosin as a non invasive biomarker in the diagnosis of breast cancer

SECONDARY OUTCOMES:
Diagnostic value of Asprosin as a biomarker in breast cancer | Baseline
  Comparing asproin and the routine markers (CEA, CA15-3) as biomarkers for diagnosis of breast cancer.

IPD SHARING:
Plan to Share IPD: No